CLINICAL TRIAL: NCT06462833
Title: The Relationship Between Health Literacy, Exercise Habits, and Medication Adherence in Postmenopausal Osteoporosis Patients
Brief Title: Health Literacy's Impact on Exercise Habits and Medication Adherence in Postmenopausal Osteoporosis
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayça Utkan Karasu, Medical Doctor, Assistant Professor, Principal Investigator, Gazi University
Other Study IDs: GaziU HL EH MA PO
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Health Literacy; Medication Adherence; Exercise; osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Medication Adherence; Motor Activity; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postmenopausal osteoporosis: Patients followed in the Physical Medicine and Rehabilitation outpatient clinic with a diagnosis of postmenopausal osteoporosis.

SUMMARY:
Postmenopausal osteoporosis is characterized by low bone mass and increased fracture risk. Treatment includes exercise, nutrition, supplements, and medications like bisphosphonates, denosumab, or hormone replacement therapy. Lifestyle changes such as quitting smoking, reducing alcohol consumption, and preventing falls are also crucial.

Despite effective treatments, adherence is low: 20-30% of patients don't start oral bisphosphonates, and 16-60% continue medications after one year. Exercise adherence rates are similarly low (14.3%-57.7%). This non-adherence imposes a significant clinical and economic burden.

Health literacy (HL)-the ability to find, understand, and use health information-is vital for managing health but is understudied in relation to osteoporosis treatment adherence. This study aims to examine the relationship between HL, exercise habits, and medication adherence in postmenopausal osteoporosis patients. Understanding these factors can lead to effective interventions, improving patient adherence and health outcomes.

The study will measure HL levels and their correlation with medication and exercise adherence, potentially informing health education programs and strategies to enhance treatment adherence. By doing so, it aims to improve health outcomes and healthcare system efficiency.

DETAILED DESCRIPTION:
Postmenopausal osteoporosis is a common bone disease characterized by low bone mass, deterioration of bone tissue microarchitecture, and an increased risk of fractures. This condition results from the imbalance between bone formation and resorption due to decreased estrogen levels. Fractures, the feared complication of osteoporosis, make this condition a significant problem both clinically and from a public health perspective. In Europe, postmenopausal osteoporosis affects approximately 22 million women and causes over 3.5 million fragility fractures annually.

Treatment options include regular exercise, healthy nutrition, calcium and vitamin D supplementation, and pharmacological treatments such as bisphosphonates, denosumab, or hormone replacement therapy. Additionally, quitting smoking, reducing alcohol consumption, and preventing falls are crucial in preventing osteoporosis and osteoporotic fractures. Despite the availability of safe and effective medications to reduce fracture risk, many patients either do not start treatment or do not adhere to it adequately. This non-adherence to treatment results in a significant clinical and economic burden. Following the prescription of medications, a substantial percentage of patients, around 20-30%, do not start taking oral bisphosphonates, and the continuation rate of osteoporosis medications over one year is reported to range from 16% to 60%. Furthermore, low levels of adherence to resistance/weight-bearing exercises (36.3%-54.4%) and physical activity (14.3%-57.7%) have been observed.

Health literacy (HL) is defined as the capacity of individuals to find, understand, evaluate, and apply health-related information to prevent diseases, develop healthy eating behaviors, and improve their health. There are limited studies on the impact of health literacy on adherence to osteoporosis treatment in postmenopausal osteoporosis patients. However, no study has investigated the effect of HL on both medical treatment adherence and exercise adherence in postmenopausal osteoporosis patients.

This study aims to investigate the relationship between health literacy, exercise habits, and medication adherence in postmenopausal osteoporosis patients. By identifying the factors leading to non-adherence to osteoporosis-preventive medications and regular exercise, effective interventions to enhance adherence to these treatments can be determined. This can result in better health outcomes for patients and increased efficiency within the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients
* Being under outpatient follow-up for osteoporosis for at least one year

Exclusion Criteria:

* Orthopedic, rheumatic, and neurological conditions that may hinder participation in exercise
* Cancer
* Refusal to participate in the study

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with postmenopausal osteoporosis and treated in the outpatient clinic for at least one year will be included in the study. Every subject meeting the criteria of inclusion is going to be included into the study via consecutive participant sampling method.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Health literacy | Patients will be evaluated once in the baseline.
  Health literacy is the capacity of individuals to find, understand, evaluate, and apply health-related information to prevent diseases, develop healthy eating behaviors, and improve their health.
  The Turkish Health Literacy Scale-32 (THLS-32) will be used to assess the health literacy levels of the patients. THLS-32 is a 32-item Likert-type scale. Scores on the scale range from 0 indicating the lowest health literacy to 50 indicating the highest health literacy.

SECONDARY OUTCOMES:
Medication adherence | Patients will be evaluated once in the baseline.
  The Medication Adherence Report Scale (MARS) will be used to assess medication adherence in patients. This scale consists of five different statements involving negative medication adherence behaviors, including deciding to skip doses, forgetting to take medication, changing the dosage, temporarily stopping medication intake, and taking less than prescribed. The total score on the MARS ranges from 5 to 25 points, with higher scores indicating better medication adherence
Physical activity | Patients will be evaluated once in the baseline.
  The International Physical Activity Questionnaire (IPAQ) was developed in 1998 for global physical activity surveillance. Since then, it has become the most widely used physical activity questionnaire. IPAQ-Short Form (IPAQ-SF) is a 7-item questionnaire that assesses the level of activity (low, moderate, high physical activity) in the past seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Utkan Karasu, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Hernlund E, Svedbom A, Ivergard M, Compston J, Cooper C, Stenmark J, McCloskey EV, Jonsson B, Kanis JA. Osteoporosis in the European Union: medical management, epidemiology and economic burden. A report prepared in collaboration with the International Osteoporosis Foundation (IOF) and the European Federation of Pharmaceutical Industry Associations (EFPIA). Arch Osteoporos. 2013;8(1):136. doi: 10.1007/s11657-013-0136-1. Epub 2013 Oct 11. PMID 24113837
- [Background] Reynolds K, Muntner P, Cheetham TC, Harrison TN, Morisky DE, Silverman S, Gold DT, Vansomphone SS, Wei R, O'Malley CD. Primary non-adherence to bisphosphonates in an integrated healthcare setting. Osteoporos Int. 2013 Sep;24(9):2509-17. doi: 10.1007/s00198-013-2326-5. Epub 2013 Apr 18. PMID 23595561
- [Background] Albrecht BM, Stalling I, Foettinger L, Recke C, Bammann K. Adherence to Lifestyle Recommendations for Bone Health in Older Adults with and without Osteoporosis: Cross-Sectional Results of the OUTDOOR ACTIVE Study. Nutrients. 2022 Jun 14;14(12):2463. doi: 10.3390/nu14122463. PMID 35745193
- [Background] Roh YH, Koh YD, Noh JH, Gong HS, Baek GH. Effect of health literacy on adherence to osteoporosis treatment among patients with distal radius fracture. Arch Osteoporos. 2017 Dec;12(1):42. doi: 10.1007/s11657-017-0337-0. Epub 2017 Apr 18. PMID 28421547